CLINICAL TRIAL: NCT01194674
Title: Microplasmin Intravitreal Administration in Participants With Uveitic Macular Edema
Acronym: MIME
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Nida Sen, M.D., Principal Investigator, NEI, National Institutes of Health Clinical Center (CC)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100186; 10-EI-0186 (Other: CNS IRB)
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Uveitis
Keywords: Microplasmin; Macular Edema; Uveitis
MeSH Terms: conditions — Uveitis; Macular Edema | interventions — microplasmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microplasmin (Experimental)
  Interventions: Drug: Microplasmin

INTERVENTIONS:
Drug: Microplasmin — Participants received an intravitreal injection of 125 µg in 100 µL of microplasmin at baseline.

SUMMARY:
The objective of this study is to investigate the safety and efficacy of microplasmin as a treatment for uveitic macular edema.

DETAILED DESCRIPTION:
Objective: Uveitis, an inflammatory condition that affects the uvea (iris, ciliary body and choroid) and adjacent structures of the eyes, is an important cause of visual loss. Most cases of uveitis, not related to an infectious agent, are thought to be autoimmune in origin and are effectively treated with medications to suppress the function of the immune system. Efforts to decrease morbidity, reduce the dose of more toxic immunosuppressive drugs, reduce the frequency of recurrences of inflammation and its sequelae are important goals in the treatment of uveitis. A frequent sequela of uveitis is macular edema. Treatment of macular edema in patients with uveitis has been a particular challenge. Current evidence from diabetic macular edema (DME) and vitreomacular traction (VMT) trials suggests that pharmacologically-induced vitreoretinal separation could be a potential treatment for macular edema associated with uveitis. Microplasmin, a truncated form of human plasmin and naturally occurring enzyme that dissolves blood clots, may be a reasonable candidate for the treatment of uveitic macular edema. The objective of this study is to investigate the safety and efficacy of microplasmin as a treatment for uveitic macular edema.

Study Population: Five participants with uveitic macular edema, with or without VMT, will be enrolled. In addition, participants must have no evidence of macular or complete posterior vitreous detachment (PVD) by Optical Coherence Tomography (OCT) or ultrasound.

Design: This Phase I-II, non-randomized, prospective, uncontrolled, single-center study will involve a one-time intravitreal injection of 125 µg in 100 µL of microplasmin. Eligible participants can receive the intravitreal injection on the same day of the baseline examination. Participants will be followed for 24 weeks post-injection.

Outcome Measures: The primary outcome measure related to the safety and tolerability of microplasmin will be assessed by the number and severity of adverse events (AEs) and systemic and ocular toxicities during the study. The secondary outcome measures related to the potential efficacy of an intravitreal injection of microplasmin for macular edema secondary to uveitis will be assessed by a change in central macular thickness from baseline measured by OCT in response to microplasmin at 4 and 12 weeks post-injection, the number of participants achieving macular or complete PVD at 4 and 12 weeks post-injection, the change of ETDRS best-corrected visual acuity (BCVA) and the change of retino-vascular leakage from baseline seen on fluorescein angiography (FA).

ELIGIBILITY:
Inclusion Criteria

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Participant has a diagnosis of uveitic macular edema that requires treatment in at least one eye (the study eye) and the uveitis in the study eye is deemed clinically quiet by the investigator.
4. Participant has no evidence of macular or complete PVD in the study eye by B-scan ultrasound and OCT.
5. Participant has visual acuity of 20/400 or better in the study eye.
6. Participant has a central macular thickness ≥ 270 microns in the study eye and loss of the normal foveal contour.
7. Participant does not have significant cataract or media opacity in the study eye that makes posterior segment visualization difficult as determined by investigator.
8. Female participants of childbearing potential must not be pregnant or breast-feeding and must have a negative serum pregnancy test at screening and throughout the study.
9. Both female participants of childbearing potential and male participants able to father a child must agree to practice two effective methods of birth control for six months following administration of study medication. Acceptable methods of birth control for this study include hormonal contraception (birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods (diaphragm, condom) with spermicide or surgical sterilization (hysterectomy, tubal ligation or vasectomy). Participants with a hysterectomy or vasectomy (or have a partner with a hysterectomy or vasectomy) are exempt from using two methods of birth control.
10. Participant is willing to comply with the study procedures and return for all study visits.

Exclusion Criteria

1. Participant has uncontrolled glaucoma, defined as intraocular pressure >30 mmHg despite treatment with anti-glaucoma medication, in the study eye.
2. Participant has lattice degeneration of the retina in the study eye deemed to be high risk by the investigator.
3. Participant has untreated retinal holes or tears, or a macular hole in the study eye.
4. Participant has a significant active ocular infection in the study eye.
5. Participant had intraocular surgery within the past 90 days or anticipates elective intraocular surgery in the study eye.
6. Participant had an injection of bevacizumab or ranibizumab within the past four weeks in the study eye.
7. Participant had an injection of triamcinolone within the past six weeks in the study eye.
8. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status that would pose a significant hazard if investigational therapy was started).
9. Participant has known anaphylaxis to sodium fluoride, or has urticaria, angioedema or an anaphylactoid response to sodium fluorescein dye that cannot be safely pre-medicated with an antihistamine and/or prednisone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Nida Sen, MD, MHSc, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gritz DC, Wong IG. Incidence and prevalence of uveitis in Northern California; the Northern California Epidemiology of Uveitis Study. Ophthalmology. 2004 Mar;111(3):491-500; discussion 500. doi: 10.1016/j.ophtha.2003.06.014. PMID 15019324
- [Background] Djalilian AR, Nussenblatt RB. Immunosuppression in uveitis. Ophthalmol Clin North Am. 2002 Sep;15(3):395-404, viii. doi: 10.1016/s0896-1549(02)00036-6. PMID 12434489
- [Background] Whitcup SM, Hikita N, Shirao M, Miyasaka M, Tamatani T, Mochizuki M, Nussenblatt RB, Chan CC. Monoclonal antibodies against CD54 (ICAM-1) and CD11a (LFA-1) prevent and inhibit endotoxin-induced uveitis. Exp Eye Res. 1995 Jun;60(6):597-601. doi: 10.1016/s0014-4835(05)80001-6. PMID 7641842
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-EI-0186.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Microplasmin
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Microplasmin
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 40.50 (17.68) [28 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Time Frame: 24 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Microplasmin
Number analyzed (Participants) | 2
Adverse Events | 4

2. Primary Outcome: Number of Severe Adverse Events
Time Frame: 24 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Microplasmin
Number analyzed (Participants) | 2
Adverse Events | 0

3. Primary Outcome: Number of Ocular Adverse Events
Description: The number of eye-related adverse events was calculated.
Time Frame: 24 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Microplasmin
Number analyzed (Participants) | 2
Adverse Events | 1

4. Primary Outcome: Number of Non-ocular Adverse Events
Description: The number of adverse events that were not eye-related was calculated.
Time Frame: 24 weeks
Measure: Number; unit: Adverse Events
Arm/Group | Microplasmin
Number analyzed (Participants) | 2
Adverse Events | 3

5. Secondary Outcome: Change in Central Macular Thickness, as Measured by Optical Coherence Tomography (OCT), at 4 Weeks vs. Baseline
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue. This protocol terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Time Frame: Baseline and 4 weeks
Population: This protocol terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Arm/Group | Microplasmin
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants Achieving Macular or Complete Posterior Vitreous Detachment (PVT) at 4 Weeks
Description: This study terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Time Frame: Baseline and 4 weeks
Population: This protocol terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Arm/Group | Microplasmin
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in ETDRS Best-corrected Visual Acuity (BCVA) at 4 Weeks vs. Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20. This study terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Time Frame: Baseline and 4 weeks
Population: This protocol terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Arm/Group | Microplasmin
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in ETDRS Best-corrected Visual Acuity (BCVA) at 12 Weeks vs. Baseline
Description: as for outcome 7
Time Frame: Baseline and 12 Weeks
Population: This protocol terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Arm/Group | Microplasmin
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Retino-vascular Leakage, as Seen on Fluorescein Angiography (FA), at 4 Weeks vs. Baseline
Description: Retino-vascular leakage was calculated after manually outlining the inner and outer borders of the subretinal fluid packet in the optical coherence tomography (OCT) images using the "Edit Segmentation" function of the Cirrus HD-OCT software. For cases in which a pigment epithelial detachment was present, the volume of the pigment epithelial detachment was included in the calculation of leakage volume. This study terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Time Frame: Baseline and 4 weeks
Population: This protocol terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Arm/Group | Microplasmin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Microplasmin
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microplasmin (N=2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes